CLINICAL TRIAL: NCT04112459
Title: Prolonged Mechanical Ventilation in Paediatric Intensive Care : An International Cross-Sectional Prevalence Study
Brief Title: LongVentKids Study
Acronym: LVK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St. Justine's Hospital (Other)
Collaborators: Réseau en Santé Respiratoire du Québec (Unknown); Fonds de la Recherche en Santé du Québec (Other Government); Women and Children's Health Research Institute, Canada (Other); Réseau mère-enfant de la francophonie (Unknown)
Responsible Party: Principal Investigator, Atsushi Kawaguchi, Postdoctoral Scholar, St. Justine's Hospital
Other Study IDs: MP-21-2019-2130
Record Dates: First submitted 2019-09-27; First posted 2019-10-02 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Prolonged Mechanical Ventilation in Pediatric Intensive Care Unit

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: prolonged mechanical ventilation — No intervention will be applied in this study

SUMMARY:
Scientific advances, population growth, lower mortality, and increasing complexity of diseases have boosted up the number of patients requiring prolonged breathing assistance with mechanical ventilators in the pediatric intensive care units (PICU) in many parts of the developed world. Previous studies also suggest that there is a small group of children who actually need such a high level of support for extended periods of time, utilizing a lot of human and technical resources. We defined children with prolonged mechanical ventilation (PMV) if they required supports with a breathing machine for more than 14 days. We propose an international point prevalence study of children requiring PMV in PICU. We will conduct the study in multiple centers in several different regions, including North and South America, Europe, and Asian countries, with a strong relationship with local physician colleagues. Practice for patients requiring PMV will be examined including the type and size of local PICU, admission and discharge policies, and patient and treatment modalities administered to such patients, types of professionals looking after patients in PMV, types of health care. We anticipate a high variability in practices suggesting a need to further standardize the management of PMV.. Specifically, as an immediate consequence, by comparing and understanding the differences in patient demographics, practice details among PICUs in regards to the background factors of local PICUs and their patients, practitioners will share their way of dealing with such patients. In that way, this study will support the need to generate guidelines and lead to patient care improvement in PICUs.

ELIGIBILITY:
Inclusion Criteria:

Patients who are ventilated >14 consecutive days (after 37 weeks postmenstrual post-conception age)*

* including for more than 6 hours per day including on InMV and NIV duration
* patient who have had and short interruptions (<48hours) of ventilation during the weaning process as the same episode of ventilation can be included.
* InMV can be administered through an endotracheal tube or a tracheostomy tube.
* NIV can be managed through a nasal, full-face, total facial mask, or helmet.
* Patient on HFNC will be included as on respiratory support if they have a proper or a nasal cannula (that allows >=1 liters/kg/min (LPM) and >4LPM).
* We define nasal oxygen supply <1 L/kg/min as non-NIV practice.

Exclusion Criteria:

* Age >18 years
* Already included in this study
* No consent if required
* Brain death
* Premature children not yet at 37 weeks gestational age.

Ages: 37 Weeks to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: All patients on invasive or non-invasive mechanical ventilation on the day of the study or patients who had been on InMV or non-invasive ventilation (NIVs) during their PICU stays will be eligible. Patients who fulfill inclusion criteria and do not meet any exclusion criteria will be considered for inclusion in the study.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2019-09-04 (Actual); Primary Completion 2021-09-03 (Estimated); Study Completion 2022-09-04 (Estimated)

PRIMARY OUTCOMES:
Prevalence of PMV | eight times during two-year study period
  number of patients meet PMV criteria devided by the number of patients admitted in PICUs on the specific data collection date and time.

SECONDARY OUTCOMES:
Patient and treatment demographics | eight times during two-year study period
  patient demographics underlying chronic disease acute disease leading to InMV or to NIV (i.e. reason of PMV) co-morbidities (Cerebral palsy, Seizure disorder, etc.) type of airway access MV mode and the days of ventilations for each mode care providers (e.g. intensivists, pediatric intensivists, anesthesiologist, paediatrician, pulmonologist) Nurse : patient ratio failed extubations or not during PMV location of patients on PMV (PICU or step down unit under PICU staff or not)
  Data from 8 study dates will be integrated into a summarized finding in the manuscript
Outcomes at 90days follow-up | 90 days from the initial data collection
  complications of mechanical ventilation mortality destination

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Jouvet, MD PhD MBA, Study Director — St. Justine's Hospital
Locations (1):
- CHU Sainte Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data sharing agreement will be mandatory to be signed between the central coordination center (CHU Sainte Justine) and the participating center.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all the data collection completed, summarized de-identified study result will be shared with the participating centers. Patient individual data will be shared between the central coordinating center and the center where PI of ancillary and posthoc study belongs.
Access Criteria: All the study protocol and CRF will be shared with the participating centers.

REFERENCES:
- [Derived] Kawaguchi A, Fernandez A, Baudin F, Chiusolo F, Lee JH, Brierley J, Colleti J Jr, Reiter K, Won Kim K, Lopez Fernandez Y, Kneyber M, Pons-Odena M, Napolitano N, Graham RJ, Kawasaki T, Garros D, Garcia Guerra G, Jouvet P; LongVentKids study group. Prevalence, management, health-care burden, and 90-day outcomes of prolonged mechanical ventilation in the paediatric intensive care unit (LongVentKids): an international, prospective, cross-sectional cohort study. Lancet Child Adolesc Health. 2025 Jan;9(1):37-46. doi: 10.1016/S2352-4642(24)00296-7. PMID 39701660